CLINICAL TRIAL: NCT04423601
Title: A Single-centre, Open, Single-dose, Self-control Study to Investigate the Effect of Itraconazole on the Pharmacokinetics of SHR6390 in Healthy Chinese Adult Subjects.
Brief Title: Effect of Itraconazole on the Pharmacokinetics of SHR6390 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR6390-I-106
Record Dates: First submitted 2020-06-07; First posted 2020-06-09 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): subjects receiving a single oral dose of SHR6390 tablets, then itraconazole capsules 200 mg/day orally with a single oral dose of SHR6390 tablets co-administered.
  Interventions: Drug: SHR6390 tablet; Drug: Itraconazole capsule

INTERVENTIONS:
Drug: SHR6390 tablet — single oral dose of SHR6390 or co-administered with itraconazole.
Drug: Itraconazole capsule — 200 mg itraconazole was administered in the morning.

SUMMARY:
The primary objective of the study is to evaluate the effect of itraconazole on pharmacokinetics of healthy Chinese adult subjects after oral administration of SHR6390 tablets. The secondary objective of the study is to evaluate the safety of SHR6390 alone and when co-administered with itraconazole. The exploratory objective of the study is to explore the effect of SHR6390 related metabolic enzymes and transporter gene polymorphisms on the pharmacokinetics of SHR6390.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent;
4. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, and body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26);

Exclusion Criteria:

1. Allergic constitution;
2. History of drug use, or drug abuse screening positive;
3. Alcoholic or often drinkers;
4. Left ventricular ejection fraction (LVEF) <50% by echocardiography;
5. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.
6. Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of SHR6390 | through study completion, an average of 32 days
  Peak Plasma Concentration (Cmax) of SHR6390
Pharmacokinetics parameter: AUC of SHR6390 | through study completion, an average of 32 days
  Area under the plasma concentration versus time curve (AUC) of SHR6390

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax of SHR6390 | through study completion, an average of 32 days
  Time of maximum observed concentration (Tmax) of SHR6390
Pharmacokinetics parameter: T1/2 of SHR6390 | through study completion, an average of 32 days
  Half time (T1/2) of SHR6390
Pharmacokinetics parameter: CL/F of SHR6390 | through study completion, an average of 32 days
  Total body clearance for extravascular administration (CL/F) of SHR6390

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided